CLINICAL TRIAL: NCT00628992
Title: Effects of Early Rehabilitation in Chronic Obstructive Pulmonary Disease Patients Under Mechanical Ventilation for Acute Respiratory Failure in Intensive Care Unit.
Brief Title: Early Rehabilitation of COPD Patients in ICU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3912
Record Dates: First submitted 2008-02-04; First posted 2008-03-05 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Acute Respiratory Failure
Keywords: COPD: chronic obstructive pulmonary disease and acute respiratory failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (4):
- 1 (Other)
  Interventions: Other: No specific intervention, standard therapy serving as a control group, passive mobilization of the legs
- 2 (Active Comparator)
  Interventions: Other: Electrical stimulation of the thigh
- 3 (Active Comparator)
  Interventions: Other: Cycloergometer training
- 4 (Active Comparator)
  Interventions: Other: Electrical stimulation of the thigh and cycloergometer training

INTERVENTIONS:
Other: No specific intervention, standard therapy serving as a control group, passive mobilization of the legs — Muscular rehabilitation of the leg
  Arms: 1
Other: Electrical stimulation of the thigh — Muscular rehabilitation of the leg
  Arms: 2
Other: Cycloergometer training — Muscular rehabilitation of the leg
  Arms: 3
Other: Electrical stimulation of the thigh and cycloergometer training — Muscular rehabilitation of the leg
  Arms: 4

SUMMARY:
Twenty per cent of the intensive care patients mechanically ventilated suffer from chronic obstructive pulmonary disease (COPD). These patients stay longer in Intensive Care which is more costly and they are more prone to nosocomial infection.In addition, they are longer bedridden and they develop muscular weakness.Prolonged inactivity results in respiratory and skeletal muscle weakness which curtails simple daily activity.The principal purpose of this study is to compare two types of muscular rehabilitation (electrical stimulation of the thigh and/or cycloergometer training) to classic passive mobilization of the leg.The second purpose is to analyse the effects of each type of rehabilitation on muscular fiber (structural and functional analysis) by muscular biopsies.Two hundred forty COPD patients admitted in the intensive care unit for acute respiratory failure will be randomized in 4: 1 fashion to receive passive mobilization of the legs(group 1, n=60), electrical stimulation of the thigh (group 2, n=60), cycloergometer training (group 3, n=60) or electrical stimulation of the thigh and cycloergometer training(group 4, n=60).The rehabilitation program will last 4 weeks with 5 sessions per week.In each group of patients, muscular biopsies will be done under local anaesthesia at the beginning and end of the rehabilitation programme and when they are discharged from the service.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years of age
* Chronic obstructive pulmonary disease
* Intubated with mechanical ventilation
* Patients without sedation or catecholamine
* 2 previous spontaneous breathing trial at 24 hour intervals with T-piece having been unsuccessful
* Conscious and cooperative state
* Ability for the patient to sit in a armchair

Exclusion Criteria:

* Non chronic obstructive pulmonary disease
* Lack of patient involvement
* Minor Patients
* Patients under guardianship
* Unconscious and non cooperative state
* Patients unable to ride in a wheelchair
* Patients not affiliated with a Social Security System
* Patients under justice safeguard
* Patients under curator ship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number day breathing without assistance during the 28-day study period | during the 28-day study period

SECONDARY OUTCOMES:
Mortality at day 28 and day 90 | Measured within the ICU stay of the patient
Length of stay in intensive care unit and hospital | Measured within the ICU stay of the patient
Clinical measurement of muscular strength in lower limbs(day 0-2 and day 28-30) | Measured within the ICU stay of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Vincent CASTELAIN, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (4):
- France (4):
  - Service de Réanimation Médicale, Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service des Explorations Fonctionnelles Respiratoires, Hôpital Civil, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service de Médecine Physique et de Réadaptation, Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service de Réanimation Médicale, Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg